CLINICAL TRIAL: NCT01142765
Title: A Phase I/IIa Sporozoite Challenge Study to Assess the Protective Efficacy of New Malaria Vaccine Candidates AdCh63 AMA1, MVA AMA1, AdCh63 MSP1, MVA MSP1, AdCh63 ME-TRAP & MVA ME-TRAP
Brief Title: Study to Assess Efficacy of New Malaria Vaccine Candidates AdCh63 AMA1, MVA AMA1, AdCh63 MSP1, MVA MSP1, AdCh63 ME-TRAP & MVA ME-TRAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Heather House, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC039
Record Dates: First submitted 2010-06-07; First posted 2010-06-11 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Malaria
Keywords: Vaccine; Safety; Immunogenicity; Protection; Sporozoite challenge
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Experimental): 1 dose of AdCh63 MSP1 and 1 dose MVA MSP1 followed by sporozoite challenge
  Interventions: Biological: AdCh63 MSP1, MVA MSP1, challenge
- Group 2 (Experimental): 1 dose of AdCh63 AMA1 and 1 dose MVA AMA1 followed by sporozoite challenge
  Interventions: Biological: AdCh63 AMA1, MVA AMA1, challenge
- Group 3 (Experimental): 1 dose of AdCh63 AMA1 and 1 dose AdCh63 MSP1 co-administered into separate arms followed by 1 dose of MVA AMA1 and 1 dose MVA MSP1 co-administered into separate arms (but the same arm as the corresponding AdCh63 vaccine) followed by sporozoite challenge
  Interventions: Biological: AdCh63 AMA1, AdCh63 MSP1, MVA AMA1, MVA MSP1, challenge
- Group 4 (Experimental): 1 dose of AdCh63 MSP1 and 1 dose AdCh63 ME-TRAP co-administered into separate arms followed by 1 dose of MVA MSP1 and 1 dose MVA ME-TRAP co-administered into separate arms (but the same arm as the corresponding AdCh63 vaccine) followed by sporozoite challenge
  Interventions: Biological: AdCh63 MSP1, AdCh63 ME-TRAP, MVA MSP1, MVA ME-TRAP, challenge
- Group 5 (Other): Non-vaccinated controls for sporozoite challenge
  Interventions: Biological: Sporozoite challenge

INTERVENTIONS:
Biological: AdCh63 MSP1, MVA MSP1, challenge — 1 dose of AdCh63 MSP1 5 x 1010 vp intramuscularly and 1 dose MVA MSP1 2.5 x 108 pfu intramuscularly 8 weeks later (range 6-12 weeks) followed by sporozoite challenge 12-28 days later
  Arms: Group 1
Biological: AdCh63 AMA1, MVA AMA1, challenge — 1 dose of AdCh63 AMA1 5 x 1010 vp intramuscularly and 1 dose MVA AMA1 2.5 x 108 pfu intramuscularly 8 weeks later (range 6-12 weeks) followed by sporozoite challenge 12-28 days later
  Arms: Group 2
Biological: AdCh63 AMA1, AdCh63 MSP1, MVA AMA1, MVA MSP1, challenge — 1 dose of AdCh63 AMA1 5 x 1010 vp intramuscularly and 1 dose AdCh63 MSP1 5 x 1010 vp intramuscularly co-administered into separate arms followed 8 weeks later (range 6-12 weeks) by 1 dose of MVA AMA1 2.5 x 108 pfu intramuscularly and 1 dose MVA MSP1 2.5 x 108 pfu intramuscularly co-administered into separate arms (but the same arm as the corresponding AdCh63 vaccine) followed by sporozoite challenge 12-28 days later.
  Arms: Group 3
Biological: AdCh63 MSP1, AdCh63 ME-TRAP, MVA MSP1, MVA ME-TRAP, challenge — 1 dose of AdCh63 MSP1 5 x 1010 vp intramuscularly and 1 dose AdCh63 ME-TRAP 5 x 1010 vp intramuscularly co-administered into separate arms followed 8 weeks later (range 6-12 weeks) by 1 dose of MVA MSP1 2.5 x 108 pfu intramuscularly and 1 dose MVA ME-TRAP 2 x 108 pfu intramuscularly co-administered into separate arms (but the same arm as the corresponding AdCh63 vaccine) followed by sporozoite challenge 12-28 days later.
  Arms: Group 4
Biological: Sporozoite challenge — Non-vaccinated controls for sporozoite challenge
  Arms: Group 5

SUMMARY:
This study aims to test the safety and efficacy of six new malaria vaccines - AdCh63 AMA1, MVA AMA1, AdCh63 MSP1, MVA MSP1, AdCh63 ME-TRAP & MVA ME-TRAP. These vaccines consist of inactivated viruses which have been modified - so they cannot reproduce (replicate) in humans, and also to include genetic material (genes) for malaria proteins which are expressed by the malaria parasite during both liver and blood stage infection. The vaccines are designed to stimulate an immune response to these malaria proteins (immunogenicity describes the nature and magnitude of this immune response) and thus provide protection against malaria infection. The protective efficacy of vaccines will be evaluated by challenging a small number of volunteers who have received the vaccines with malaria infection from the bites of infected mosquitos(sporozoite challenge).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For female volunteers, willingness to practice continuous effective contraception for the duration of the study.
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

* History of clinical P. falciparum malaria
* Travel to a malaria endemic region during the study period or within the preceding six months with a risk of malaria exposure.
* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* Pregnancy, lactation or intention to become pregnant during the study
* Contraindication to both anti-malarial drugs; Riamet & chloroquine

  * Concomitant use with other drugs known to cause QT-interval prolongation (e.g. macrolides, quinolones, amiodarone etc)
  * History of epilepsy
* History of arrhythmia or prolonged QT interval.
* Family history for sudden cardiac death.
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system 107
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine e.g. egg products, Kathon.
* History of clinically significant contact dermatitis
* Any history of anaphylaxis post vaccination
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition that may affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Any clinically significant abnormal finding on biochemistry or haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of vaccine | Up to 18 months
  To assess if volunteers who receive the novel vaccine candidates; AdCh63 MSP1, MVA MSP1, AdCh63 AMA1, MVA AMA1, AdCh63 ME-TRAP and MVA ME-TRAP in heterologous prime boost regimens are protected wholly or partially against malaria infection in a sporozoite challenge model. This will be determined by noting the number of subjects who develop malaria infection and the time in hours between exposure and parasitaemia as detected by thick-film blood smear compared with controls.
  To assess the safety of the immunisation regimens alone and during co-administration.

SECONDARY OUTCOMES:
Immunogenicity of vaccine | Up to 18 months
  To assess immunogenicity of the vaccine regimes by measuring IFN-γ ELISPOT, flow cytometry and antibody responses to MSP1, AMA1 and ME-TRAP antigens before and after malaria infection. If there is evidence of partial or complete protection, we will explore immunological correlates of protective immunity.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, D.Phil, FRCP, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Hospital for Tropical Diseases Mortimer Market, London
  - Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford
  - Wellcome Trust Clinical Research Facility, University of Southampton, Southampton